CLINICAL TRIAL: NCT02206620
Title: Effects of Cholinergic Augmentation on Measures of Balance and Gait
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Principal Investigator, John G. Nutt, M.D., Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9437
Record Dates: First submitted 2014-07-29; First posted 2014-08-01 (Estimated); Results first posted 2019-11-14 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Donepezil (Experimental): Donepezil 5 mg per day for week 1-3 or 12-14. 10 mg/day for weeks 4-6 or 14-18, if tolerated.
  Interventions: Drug: Donepezil
- Placebo (Placebo Comparator): Placebo 5 mg per day for week 1-3 or 12-14. 10 mg/day for weeks 4-6 or 14-18, if tolerated.
  Interventions: Drug: Donepezil

INTERVENTIONS:
Drug: Donepezil
  Other Names: Aricept

SUMMARY:
This study will compare the effects of placebo and donepezil, a drug that helps conserve concentrations of the neurotransmitter, acetylcholine, on measures of balance and gait in subjects with Parkinson's disease (PD). This study is a double-blind, placebo controlled, cross-over randomized clinical trial. Short-latency afferent inhibition (SAI), a physiological index of cholinergic function will be measured to determine if the deficits in balance and gait correlate with abnormalities of the SAI and if SAI is altered by donepezil as a measure of drug efficacy. Cognitive tests like the Attention Network Test (ANT) will be administered to determine if changes in gait and balance are mediated by changes in attention.

The results of this study will be the most direct test of the hypothesized role of cholinergic neurons and the neurotransmitter, acetylcholine in terms of gait and balance. The study is exploratory because it is not known whether donepezil will affect gait, balance or attention, nor which measures of gait, balance or attention will be sensitive to drug manipulation. The study's immediate goal is to determine the potential utility of cholinergic manipulation as a strategy for preventing or treating balance and gait dysfunction in PD. The findings of this trial are intended to lead to more sharply focused questions about the role of cholinergic neurons in balance and gait and eventually to Phase II B trials to determine clinical utility of cholinergic manipulation to prevent falls and improve mobility.

ELIGIBILITY:
Inclusion Criteria:

* 30 years old or older
* Diagnosis of idiopathic Parkinson's disease
* Stand unassisted (without use of an assistance device) and walk continuously for at least 2 minutes.

Exclusion Criteria:

* musculoskeletal disorders that affect standing and walking
* Uncorrected vision disturbance
* Vestibular problems
* Major depression
* Hallucinations or other psychiatric disturbances
* Tachycardia
* Bradycardia
* Arrhythmias
* Peptic ulcer disease
* Use of anticholinergics
* Use of cholinesterase inhibitors
* Use of bladder antispasmodics
* Use of tricyclic antidepressants

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Nutt, M.D., Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mancini M, Fling BW, Gendreau A, Lapidus J, Horak FB, Chung K, Nutt JG. Effect of augmenting cholinergic function on gait and balance. BMC Neurol. 2015 Dec 23;15:264. doi: 10.1186/s12883-015-0523-x. PMID 26697847
- See also: The Michael J. Fox Foundation "Fox Trial Finder" Study Listing — https://foxtrialfinder.michaeljfox.org/trial/3851/

RESULTS

PARTICIPANT FLOW:
Groups:
- Donepezil, Then Placebo: Donepezil 5 mg per day for weeks 1-3. 10 mg/day for weeks 4-6. Then 6 week washout followed by 6 weeks of placebo. Placebo (identical appearing capsules), two capsules per day for 2 weeks and four capsules per day for the following 2 weeks.
- Placebo, Then Donepezil: Placebo (identical appearing capsules), two capsules per day for weeks 1-3 and four capsules per day for 4-6 weeks followed by washout for 6 weeks and then crossover to donepezil for six weeks. Donepezil 5 mg per day for 2 weeks, then 10 mg/day for the following 2 weeks.
Period: Phase I - First Intervention (6 Weeks)
Arm/Group | Donepezil, Then Placebo | Placebo, Then Donepezil
Started | 22 | 27
Completed | 21 | 26
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Washout (6 Weeks)
Arm/Group | Donepezil, Then Placebo | Placebo, Then Donepezil
Started | 21 | 26
Completed | 21 | 26
Not Completed | 0 | 0
Period: Phase II - Second Intervention (6 Weeks)
Arm/Group | Donepezil, Then Placebo | Placebo, Then Donepezil
Started | 21 | 26
Completed | 21 | 24
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Donepezil was taken for 3 weeks at 5mg/day (1 tablet/day) and then increased to 10mg/day (2 tablets/day) for another 3 weeks. The same was done for the placebo (1 tablet for the first 3 weeks, then 2 tablets for the following 3 weeks). There was a washout period of 6 weeks between the interventions. Participants were randomized to start with donepezil or placebo.
Arm/Group | All Study Participants
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 35
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Disease Duration [Mean (Standard Deviation); unit: years] | 7 (5)
MoCA [Mean (Standard Deviation); unit: scores on a scale] — Montreal Cognitive Assessment: overall cognition. Scale from 0 to 30. 30 represents intact cognitive status
  scores on a scale | 26 (3)
MDS-UPDRS Part III [Mean (Standard Deviation); unit: units on a scale] — Unified Parkinson's Disease Rating Scale (UPDRS), Movement Disorders Society (MDS) revised. Participants are rated on a variety of motor functions in a series of subscales. Subscale scores range from 0 to 4. The sub scales are summed to get the total score. The total score minimum score is 0 and the maximum score is 132. Higher values represent further disease progression.
  units on a scale | 43 (12)

OUTCOME MEASURES:

1. Primary Outcome: Delta Medio-lateral Postural Sway Range (Foam)
Description: Increased body sway while standing may be markers for increased risk of falling in Parkinson's disease. Sway was measured with an inertial sensor attached to the waist. Participants did this task on a foam pad. We reported the delta in the donepezil and placebo phases [post-donepezil - pre-donepezil for the donepezil phase, and post-placebo - pre-placebo for the placebo phase].
Time Frame: Six weeks
Measure: Mean (Standard Deviation); unit: m/s^2
Groups:
- Donepezil: Donepezil 5 mg per day for week 1-3 or 12-14. 10 mg/day for weeks 4-6 or 14-18, if tolerated.
  Donepezil
- Placebo: Placebo 5 mg per day for week 1-3 or 12-14. 10 mg/day for weeks 4-6 or 14-18, if tolerated.
  Donepezil
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 49 | 49
m/s^2 | 0.007 (0.045) | -0.004 (0.028)

2. Primary Outcome: Delta of the Variability of Stride Time While Walking
Description: Variability in stride time time and an increase with dual tasking is another marker for increased fall risk in Parkinson's disease. Stride time variability was measured with inertial sensors attached to both feet. The delta for each phase is reported [post-donepezil - pre-donepezil for the donepezil phase, and post-placebo - pre-placebo for the placebo phase].
Time Frame: Six weeks
Population: Variability of stride time was calculated from the stride time time-series as the coefficient of variation (CV, 100 multiplied by the SD of the stride times divided by the mean of each subject's stride times)
Measure: Mean (Standard Deviation); unit: percentage of gait cycle time
Groups:
- Donepezil: Donepezil 5 mg per day for week 1-3. 10 mg/day for weeks 4-6. Then 6 week washout followed by 6 weeks of placebo.
- Placebo: Placebo (identical appearing capsules), two capsules per day for week 1-3 and four capsules per day for 4-6 weeks followed by washout for 6 weeks and then crossover to donepezil for six weeks.
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 49 | 49
percentage of gait cycle time | -0.32 (4.07) | -0.038 (3.98)

3. Secondary Outcome: Short-latency Afferent Inhibition is a Marker of Cortical Cholinergic Activity
Description: Short-latency afferent inhibition (SAI) by a peripheral stimulation is a transcranial magnetic stimulation method to evaluate cortical cholinergic activity. Short-latency afferent Inhibition will be used to determine if our subjects with Parkinson's disease have evidence of reduced cholinergic tone which correlates with their measures of postural and gait instability. We report the SAI at the end of each phase (post-placebo phase and post-donepezil phase). SAI is reported in motor-evoked potential (MEP).
Time Frame: Six weeks
Population: The average and standard deviation (SD) of the SAI at the end of each treatment is reported
Measure: Mean (Standard Deviation); unit: percentage of the unconditioned MEP
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 49 | 49
percentage of the unconditioned MEP | 72.5 (26.9) | 74.3 (23.8)

4. Secondary Outcome: Attention Network Test
Description: Attention Network Test (ANT) is 15 minute computerized test or reaction times with various cues and targets designed to assess alerting, orienting and executive control of attention. Deficits of attention are related to fall risk and may be affected by donepezil.
  The delta of the Orienting Network Efficiency is reported for each phase (pre- and post-donepezil phase and pre- and post-placebo phase).
  Details: In accordance with Fan et al. (2002), the subtraction method was applied to isolate the efficiency of the three attentional networks as follows: for the alerting network efficiency: mean RT NC trials - mean RT DC trials; for the orienting network efficiency: mean RT CC trials - mean RT SC trials; and for the executive network efficiency: mean RT I trials - mean RT C trials. For both the alerting and orienting effects, higher subtraction scores indicate greater efficiency; by contrast, the more efficient the executive network is, the lower the subtraction score.
Time Frame: Six weeks
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 49 | 49
ms | -19.5 (16.3) | -5.1 (5.9)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected through study completion, an average of 18 weeks.
Description: Adverse Events were systematically collected by phone call every week. Study clinicians recorded adverse events and reported to the IRB unexpected or serious adverse events. An independent neurologist reviewed the reported adverse events each six months and made recommendations to the trial leadership as well as the IRB about advisability of continuation of the trial.
  The adverse events are reported below per intervention for each Arm/Group of the study.
Groups:
- Donepezil, Then Placebo (Phase I): Participants took a donepezil 5mg tablet each day for 3 weeks, then increased the dose to 10mg (2 tablets each day) for 3 weeks. (This was followed by 6 weeks of a washout period and then taking the placebo in the same format -- 3 weeks of one tablet, followed by 3 weeks of 2 tablets to replicate the dosage increase.)
- Placebo, Then Donepezil (Phase I): Participants took the placebo at one tablet each day for 3 weeks, then increased the dosage to 2 tablets each day for 3 weeks. (This was followed by 6 weeks of a washout period and then taking donepezil in the same format -- donepezil 5mg tablet each day for 3 weeks, followed by 3 weeks of an increased dose of 10mg (2 tablets each day).)
- Donepezil, Then Placebo (Washout): There were 6 weeks of a washout period after participants had taken donepezil for 6 weeks.
- Placebo, Then Donepezil (Washout): There were 6 weeks of a washout period after participants had taken the placebo for 6 weeks.
- Donepezil, Then Placebo (Phase II): After the washout period, participants took the placebo in the same format as the donepezil -- 3 weeks of one tablet, followed by 3 weeks of 2 tablets to replicate the dosage increase.
- Placebo, Then Donepezil (Phase II): Then participants took donepezil in the same formats the placebo -- the donepezil 5mg tablet each day for 3 weeks, followed by 3 weeks of an increased dose of 10mg (2 tablets each day).
Arm/Group | Donepezil, Then Placebo (Phase I) | Placebo, Then Donepezil (Phase I) | Donepezil, Then Placebo (Washout) | Placebo, Then Donepezil (Washout) | Donepezil, Then Placebo (Phase II) | Placebo, Then Donepezil (Phase II)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/27 | 0/21 | 0/26 | 0/21 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/27 | 0/21 | 1/26 | 0/21 | 0/26
Other Adverse Events (participants affected / at risk) | 18/22 | 18/27 | 5/21 | 8/26 | 4/21 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Donepezil, Then Placebo (Phase I) (N=22) | Placebo, Then Donepezil (Phase I) (N=27) | Donepezil, Then Placebo (Washout) (N=21) | Placebo, Then Donepezil (Washout) (N=26) | Donepezil, Then Placebo (Phase II) (N=21) | Placebo, Then Donepezil (Phase II) (N=26)
Pulmonary Embolus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Donepezil, Then Placebo (Phase I) (N=22) | Placebo, Then Donepezil (Phase I) (N=27) | Donepezil, Then Placebo (Washout) (N=21) | Placebo, Then Donepezil (Washout) (N=26) | Donepezil, Then Placebo (Phase II) (N=21) | Placebo, Then Donepezil (Phase II) (N=26)
Anorexia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 6 | 2 | 0 | 1 | 2 | 8
Diarrhea (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 3
Constipation (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 2
Abdominal Pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 1
Insomnia (General disorders) | 3 | 5 | 1 | 1 | 1 | 6
Vivid Dreams (General disorders) | 2 | 2 | 0 | 0 | 0 | 2
Fatigue (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0 | 0 | 2 | 3
Muscle Cramps (Musculoskeletal and connective tissue disorders) | 3 | 3 | 2 | 0 | 1 | 5
Light Headedness (General disorders) | 3 | 4 | 0 | 2 | 1 | 3
Headache (General disorders) | 2 | 0 | 0 | 0 | 0 | 0
Hallucinations (General disorders) | 2 | 0 | 1 | 1 | 1 | 1
Memory Disturbances (General disorders) | 1 | 2 | 0 | 1 | 0 | 0
Increased Saliva (General disorders) | 1 | 1 | 0 | 0 | 0 | 0
Decreased Saliva (General disorders) | 0 | 2 | 0 | 0 | 0 | 0
Urinary Frequency (Renal and urinary disorders) | 2 | 4 | 0 | 0 | 0 | 4
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 0 | 1 | 0 | 0
Other (General disorders) | 4 | 5 | 2 | 2 | 1 | 7 — other adverse events consisting of Irregular Heartbeat, Pain, Weakness, Anxiety, Excessive Sweating, Trouble Swallowing, Infection, Rash, Food Poisoning, Impulse Control, Increased Freezing of Gait, etc

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-15): https://cdn.clinicaltrials.gov/large-docs/20/NCT02206620/Prot_SAP_000.pdf